CLINICAL TRIAL: NCT06882109
Title: The 5-in-2 Ankle Block for Outpatient Foot Surgery: the FIT Block Descriptive Study
Brief Title: The 5-in-2 Ankle Block for Outpatient Foot Surgery: the FIT Block Study
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Principal Investigator, CAPDEVILA Xavier, (MD, PhD) Principal investigator, University Hospital, Montpellier
Other Study IDs: IORG0010765; CER-2024-XC01 (Other: Comité d'Ethique pour la Recherche Saint Jean (CER Saint-Jean))
Record Dates: First submitted 2025-02-25; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Foot Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Five-in-two ankle block — The FIT block is a new approach for regional anesthetic block of the ankle. We use an optimized ultrasound guided approach for the FIT Block, based on optimal nerve anatomical locations. A one puncture proximal approach for the fibular nerves is used, while maintaining the benefit of preserved extrinsic motricity. Another one puncture approaches the sural nerve laterally, after the block of the tibial nerve during the same puncture and then the subcutaneous infiltration of the saphenous nerve. An anatomical proof of concept study has been done before the exploratory clinical study.
  These approaches permit a surgical anesthetic block for foot surgery using 2 punctures (instead of 5) with a single patient's body position, compatible with sedation.

SUMMARY:
Hallux valgus surgery is known as a painful surgery. Qualitative pain management is the key to successful early recovery and rehabilitation.

Popliteal sciatic nerve block is widely used but at risk of falling due to prolonged motor blockade and foot drop. Ankle block is recognized as a good regional anesthesia technique but requires five skin punctures.

FIT block might be a good alternative, aiming to provide an optimal anesthetic block, good postoperative analgesia without motor blockade (calf muscles) and necessitating only two skin punctures.

The purpose of this study is to describe the technique and the efficacy and safety of the FIT block for outpatient foot surgery

DETAILED DESCRIPTION:
Foot surgery is frequently performed using regional anesthesia (RA). The ultrasound guided popliteal sciatic nerve block seems the gold standart technique. Improved ultrasound resolution and the development of early rehabilitation in outpatient surgery have led to the development of more distal RA techniques, at the ankle.

The ankle blocks are well described and provide similar anesthetic quality and surgical comfort than the popliteal sciatic nerve block. However, it has been reported that successful surgical anesthesia with ankle block was not reached in 14% to 16% of patients scheduled for hallux valgus surgery. Interestingly, these distal blocks preserve extrinsic motor function of the foot, enabling the patient to ambulate while minimizing the risk of falling.

Distal blocks using repeated punctures close to the periostum are painful during the RA performance. Sensitivity is greater at limbs extremities, as evidenced by Penfield's homonculus and the size of the brain surface devoted to extremities. As a result, it is frequently necessary to sedate the patient during the regional anesthesia procedure. The position of the ankle tourniquet may also require sedation if the surgery is to be prolonged.

For foot surgery under ankle blocks, it is necessary to anesthetize all distal branches of the sciatic nerve, i.e. the superficial and deep fibular nerves, the tibial nerve and the sural nerve. The saphenous nerve, coming from the lumbar plexus, is anesthetized with an ankle skin infiltration.

In the classical approaches, the tibial nerve is blocked at the medial aspect of the ankle, in the medial retro-malleolar region, posterior to tibial vessels. The sural nerve is blocked superficially in the lateral retro-malleolar region, between the calcaneal tendon and the lateral malleolus. The deep fibular nerve is located on the anterior surface of the instep, next to the periosteum, particularly painful when encountered by the needle. The superficial fibular nerve is located on the anterolateral aspect of the leg, where it is already divided into its two distal branches. Sometimes not visualized on ultrasound, these branches can be blocked by subcutaneous infiltration. This presents a risk of failure due to the anatomical variability of their emergence, explaining the risk of sensory blockade failure, as well as a theoretical risk of accidental injury during infiltration.

Optimized ultrasound guided approach for the FIT Block will be used, based on optimal nerve anatomical locations. A one puncture proximal approach for the fibular nerves is used, while maintaining the benefit of preserved extrinsic motricity. Another one puncture approaches the sural nerve laterally, after the block of the tibial nerve during the same puncture and then the subcutaneous infiltration of the saphenous nerve. An anatomical proof of concept study has been done before the exploratory clinical study.

These approaches permit a surgical anesthetic block for foot surgery using 2 punctures (instead of 5) with a single patient's body position, compatible with sedation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years old
* Scheduled for outpatient foot surgery and undergoing a FIT-block as regional anesthesia

Exclusion Criteria:

* Severe coagulopathy
* Peripheral neuropathy or chronic pain syndrome
* Infection or injury at the needle entry points
* Allergy or contraindications to study drugs
* Pregnancy or breastfeeding woman
* Inability to participate in pain scoring scales

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with FIT-Block for outpatient foot surgery
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Complete motor and sensory blocks | From 30 min after regional anesthesia to discharge from the operating room
  Complete motor and sensory blocks required for surgery under exclusive regional anesthesia by 5-in-2 ankle block

SECONDARY OUTCOMES:
Duration of the 5-in-2 ankle block | From 30 min after regional anesthesia to 24 hours after surgery
  Delay before the resolution of motor and sensory blocks
Pain intensity | From leaving the operating room to 24 hours after surgery
  Measured by Visual Analogue Scale (VAS) at rest and during movement from 0 (no pain) to 10 (worst pain).
Morphine sulfate consumption | From leaving the operating room to 24 hours after surgery
  The total morphine sulfate consumption from the operating room discharge to 24 hours after surgery
Patient satisfaction | The day after surgery (24 hours)
  Assessed by EVAN-LR questionnaire (Evaluation du Vécu de l'Anesthésie LocoRégionale) from 0 (worst satisfaction) to 10 (best satisfaction).

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Deffontis, MD, Principal Investigator — University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: No